CLINICAL TRIAL: NCT02682160
Title: Pilot Study to Evaluate the Evolution of Daily Protein Intake in Obese Patients With Recent Bariatric Surgery, Using the Software Protein Assistant.
Brief Title: Pilot Study to Evaluate Daily Protein's Intake Following Bariatric Surgery by Using the Software Protein Assistant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14 7310 02
Record Dates: First submitted 2016-02-05; First posted 2016-02-15 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of Protein Assistant (Other): patients can use the Protein Assistant during 2 months to evaluate the quantity of protein's intake.
  Interventions: Other: use of Protein Assistant

INTERVENTIONS:
Other: use of Protein Assistant — The patient has to complete a dietary record every 2 weeks during 2 months (month 2 and 3 after surgery). The aim is to intake 60g per day. If the aim is not reached, Protein assistant suggests qualitative and/or quantitative solutions.

SUMMARY:
The aim of this study is to evaluate the effect of the use of Protein Assistant on the daily protein intake in obese patients who underwent a bariatric surgery (in the 3 months following surgery).

DETAILED DESCRIPTION:
After a bariatric surgery, food intake is reduced. Patients should favor proteins to avoid loss of muscles. The guidelines recommend a minimal protein's intake of 60g per day. But this goal is achieved only for 55 to 60 % patients 4 months after surgery and 50 à 65 % patients at one year.

Protein assistant is a software which can calculate the amount of proteins eaten per day and can propose solutions if the intake is insufficient.

The main objective of this study is to evaluate the effect of the use of Protein Assistant on the daily protein intake in obese patients who underwent a bariatric surgery (in the 3 months following surgery).

Protein Assistant is suggested 1 month after bariatric surgery on a digital tablet. The patient is educated to use Protein Assistant. The patient has to complete a dietary record every 2 weeks during 2 months. The aim is to intake 60g per day. If the aim is not reached, Protein assistant suggests qualitative and/or quantitative solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a bariatric surgery a month +/- one week ago
* Able to use a digital tablet
* With internet access at home
* Accepting modalities of formation and of digital tablet lending
* When the average of protein intake is under 60g/j on a 3 days dietary record, one month after bariatric surgery

Exclusion Criteria:

* Lack of understanding of the use of a digital tablet
* Under the protection of justice
* Person participating to another trial
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the evolution of the average of protein's intake in grams/day (calculated on a 3 day's dietary record) between the first record and the last one (3 months after surgery) | 3 months after surgery

SECONDARY OUTCOMES:
the effect of Protein Assitant's use : evaluation of the % of patients reaching the goal of 60g per day of protein's intake 3 months after surgery and at each dietary record. | 3 months after surgery
patient's satisfaction | 3 months after surgery
  measured by the % of questionnaire response

CONTACTS AND LOCATIONS:
Overall Officials: Ana Estrade, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Estrade A, Montastier E, Turnin MC, Buisson JC, du Rieu MC, Tuyeras G, Hernandez G, Berard E, Ritz P. An Application May Help Improve Protein Consumption after Bariatric Surgery. Obes Surg. 2019 Jun;29(6):1982-1983. doi: 10.1007/s11695-019-03816-5. PMID 30880355